CLINICAL TRIAL: NCT01881789
Title: Phase 1b/2, Multicenter, Open-label Study of Oprozomib and Dexamethasone, in Combination With Lenalidomide or Oral Cyclophosphamide in Patients With Newly Diagnosed Multiple Myeloma
Brief Title: Oprozomib and Dexamethasone,in Combination With Lenalidomide or Oral Cyclophosphamide to Treat Newly Diagnosed Multiple Myeloma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: A program evaluation identified that the safety profile and pharmacokinetic (PK) characteristics of the formulation used in all oprozomib studies required further optimization and thus enrollment in OPZ003 was halted during dose-escalation.
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: OPZ003; 20130410 (Other: Amgen Study ID)
Record Dates: First submitted 2013-06-13; First posted 2013-06-20 (Estimated); Results first posted 2021-03-03 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Multiple Myeloma
Keywords: multiple myeloma; proteasome inhibitor; oprozomib; orpozomib tablets
MeSH Terms: conditions — Multiple Myeloma | interventions — ONX 0912; Lenalidomide; Dexamethasone; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Oprozomib 150 mg 5/14 + Lenalidomide + Dexamethasone (Experimental): Participants received oprozomib 150 mg once daily on days 1 to 5 and days 15 to 19 (5/14 schedule) of each 28-day treatment cycle, in combination with lenalidomide 25 mg on days 1 through 21 and dexamethasone 20 mg/day on days 1, 2, 8, 9, 15, 16, 22, and 23, until progression of disease, unacceptable toxicity, or for 24 cycles, whichever occurred first. After completing 24 cycles of treatment, participants with stable disease or better could have continued on oprozomib with or without dexamethasone pretreatment.
  Interventions: Drug: Oprozomib; Drug: Lenalidomide; Drug: Dexamethasone
- Oprozomib 180 mg 5/14 + Lenalidomide + Dexamethasone (Experimental): Participants received oprozomib 180 mg once daily on days 1 to 5 and days 15 to 19 (5/14 schedule) of each 28-day treatment cycle, in combination with lenalidomide 25 mg on days 1 through 21 and dexamethasone 20 mg/day on days 1, 2, 8, 9, 15, 16, 22, and 23, until progression of disease, unacceptable toxicity, or for 24 cycles, whichever occurred first. After completing 24 cycles of treatment, participants with stable disease or better could have continued on oprozomib with or without dexamethasone pretreatment.
  Interventions: Drug: Oprozomib; Drug: Lenalidomide; Drug: Dexamethasone
- Oprozomib 210 mg 5/14 + Lenalidomide + Dexamethasone (Experimental): Participants received oprozomib 210 mg once daily on days 1 to 5 and days 15 to 19 (5/14 schedule) of each 28-day treatment cycle, in combination with lenalidomide 25 mg on days 1 through 21 and dexamethasone 20 mg/day on days 1, 2, 8, 9, 15, 16, 22, and 23, until progression of disease, unacceptable toxicity, or for 24 cycles, whichever occurred first. After completing 24 cycles of treatment, participants with stable disease or better could have continued on oprozomib with or without dexamethasone pretreatment.
  Interventions: Drug: Oprozomib; Drug: Lenalidomide; Drug: Dexamethasone
- Oprozomib 210 mg 2/7 + Lenalidomide + Dexamethasone (Experimental): Participants received oprozomib 210 mg once daily on days 1, 2, 8, 9, 15, 16, 22, and 23 (2/7 schedule) of each 28-day treatment cycle, in combination with lenalidomide 25 mg on days 1 through 21 and dexamethasone 20 mg/day on days 1, 2, 8, 9, 15, 16, 22, and 23, until progression of disease, unacceptable toxicity, or for 24 cycles, whichever occurred first. After completing 24 cycles of treatment, participants with stable disease or better could have continued on oprozomib with or without dexamethasone pretreatment.
  Interventions: Drug: Oprozomib; Drug: Lenalidomide; Drug: Dexamethasone
- Oprozomib 240 mg 2/7 + Lenalidomide + Dexamethasone (Experimental): Participants received oprozomib 240 mg once daily on days 1, 2, 8, 9, 15, 16, 22, and 23 (2/7 schedule) of each 28-day treatment cycle, in combination with lenalidomide 25 mg on days 1 through 21 and dexamethasone 20 mg/day on days 1, 2, 8, 9, 15, 16, 22, and 23, until progression of disease, unacceptable toxicity, or for 24 cycles, whichever occurred first. After completing 24 cycles of treatment, participants with stable disease or better could have continued on oprozomib with or without dexamethasone pretreatment.
  Interventions: Drug: Oprozomib; Drug: Lenalidomide; Drug: Dexamethasone
- Oprozomib 210 mg 2/7 + Cyclophosphamide + Dexamethasone (Experimental): Participants received oprozomib 210 mg once daily on days 1, 2, 8, 9, 15, 16, 22, and 23 (2/7 schedule) of each 28-day treatment cycle, in combination with oral cyclophosphamide 300 mg/m² on days 1, 8, and 15 and dexamethasone 20 mg/day on days 1, 2, 8, 9, 15, 16, 22, and 23, until progression of disease, unacceptable toxicity, or for 8 cycles, whichever occurred first. After completing 8 cycles of treatment, participants with stable disease or better were to continue on oprozomib with dexamethasone premedication for a total of 24 cycles or until progression of disease or unacceptable toxicity. After completing 24 cycles of treatment, participants without evidence of disease progression could have continued on oprozomib with or without dexamethasone pretreatment.
  Interventions: Drug: Oprozomib; Drug: Dexamethasone; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Oprozomib — Extended release (ER) tablets administered orally
  Other Names: Oprozomib ER tablets
Drug: Lenalidomide — Administered orally at a dose of 25 mg on days 1 through 21 of each 28-day cycle for a maximum of 24 cycles.
  Other Names: Revlimid
  Arms: Oprozomib 150 mg 5/14 + Lenalidomide + Dexamethasone; Oprozomib 180 mg 5/14 + Lenalidomide + Dexamethasone; Oprozomib 210 mg 2/7 + Lenalidomide + Dexamethasone; Oprozomib 210 mg 5/14 + Lenalidomide + Dexamethasone; Oprozomib 240 mg 2/7 + Lenalidomide + Dexamethasone
Drug: Dexamethasone — Administered at 20 mg, orally, on days 1, 2, 8, 9, 15, 16, 22, and 23 of each 28-day cycle. After the first cycle the dose may be decreased to 10 mg/day in participants > 75 years of age, at the discretion of the investigator.
Drug: Cyclophosphamide — Administered orally at 300 mg/m² (up to a maximum of 600 mg) on days 1, 8, and 15 of each 28-day cycle for a maximum of 8 cycles of therapy (approximately 8 months).
  Other Names: Cytoxan
  Arms: Oprozomib 210 mg 2/7 + Cyclophosphamide + Dexamethasone

SUMMARY:
The primary objectives of this study included the following:

Phase 1b:

* To establish the maximum tolerated dose (MTD) of oprozomib given in combination with lenalidomide and dexamethasone (ORd) or with cyclophosphamide and dexamethasone (OCyd)
* To evaluate the safety and tolerability of oprozomib and dexamethasone administered in combination with lenalidomide or oral cyclophosphamide

Phase 2:

* To estimate the antitumor activity of each combination regimen, as measured by overall response rate (ORR) and complete response rate (CRR)
* To evaluate the safety and tolerability of each combination regimens, as assessed by the type, incidence, severity and seriousness of adverse events, and abnormalities in selected laboratory analytes

DETAILED DESCRIPTION:
Phase 1b used a standard 3 + 3 dose-escalation scheme to determine the MTD. For each combination regimen, oprozomib doses were to be escalated in sequential cohorts of 3 participants with expansion to up to 6 participants if a dose-limiting toxicity (DLT) was observed in 1 of the first 3 participants. The doses of lenalidomide, cyclophosphamide, and dexamethasone were to remain fixed in all dose cohorts.

The phase 2 portion of the study was to include up to 35 additional participants in each of the 2 combination regimens, treated at the recommended phase 2 dose (RP2D) of oprozomib that was identified during the phase 1b portion of the study in order to better characterize safety and tolerability, and antimyeloma activity.

This study was stopped by sponsor decision during the dose escalation in phase 1b prior to initiation of phase 2.

ELIGIBILITY:
Key Inclusion Criteria:

* Newly diagnosed, symptomatic multiple myeloma patients for whom treatment is indicated per the National Comprehensive Cancer Network (NCCN) guidelines, and for whom a hematopoietic stem cell transplant is not planned or scheduled during the study or are considered ineligible for hematopoietic stem cell transplant, with measurable disease
* Creatinine clearance of ≥ 50 mL/min (measured or calculated using the Cockcroft and Gault formula)

Key Exclusion Criteria:

* Any prior systemic antimyeloma therapy except oral steroids (dexamethasone up to a total dose of 160 mg or equivalent within 14 days prior to the first dose of study treatment). Use of topical or inhaled steroids is acceptable
* Radiation therapy within 2 weeks prior to first dose
* Major surgery within 3 weeks prior to first dose
* Active infection requiring systemic antibiotics, antivirals, or antifungals within 2 weeks prior to first dose
* Clinical significant gastrointestinal bleeding in the 6 months prior to Cycle 1 Day 1 (C1D1) first dose
* Significant neuropathy (Grade 3, Grade 4, or Grade 2 with pain) at the time of first dose
* Other malignancy within the past 3 years except those considered cured by surgical resection including some cases of: with the exception of adequately treated basal or squamous cell carcinoma of the skin, squamous cell skin cancer, thyroid cancer, carcinoma in situ of the breast or cervix, carcinoma in situ of the breast, prostate cancer with Gleason Score 6 or less with stable prostate specific antigen levels, or cancer considered cured by surgical resection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2013-10-28 (Actual); Primary Completion 2019-09-23 (Actual); Study Completion 2019-09-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (14):
- United States (14):
  - Clearview Cancer Institute, Huntsville, Alabama
  - Providence St. Joseph's Hospital, Burbank, California
  - David Geffen School of Medicine at UCLA, Los Angeles, California
  - Monterey Bay Oncology Corp DBA Pacific Cancer Care, Salinas, California
  - Colorado Blood Cancer Institute, Denver, Colorado
  - H. Lee Moffit Cancer Center & Research Institute, Tampa, Florida
  - University of Chicago Medical Center, Chicago, Illinois
  - Indiana University Health Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Center for Cancer & Blood Disorders, Bethesda, Maryland
  - The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - University of Texas M.D. Anderson Cancer Center, Houston, Texas
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Froedtert Hospital and the Medical College of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 17 study centers in the United States. Twenty-two participants were enrolled, however one participant discontinued before being assigned to a treatment cohort.
  Enrollment was halted during dose-escalation and Phase 2 was not conducted.
Pre-assignment Details: In the Phase 1b portion of the study participants were enrolled sequentially using a standard 3 + 3 dose escalation schema.
  The final planned analysis for efficacy was performed using a data cut-off date of 18 July 2016, at which time 3 participants remained on treatment. The final analysis of safety was conducted after all participants had discontinued treatment (23 September 2019).
Groups:
- Oprozomib 210 mg 5/14 + Lenalidomide + Dexamethasone: Participants received oprozomib 210 mg once daily on days 1 to 5 and days 15 to 19 (5/14 schedule) of each 28-day treatment cycle, in combination with lenalidomide 25 mg on days 1 through 21 and dexamethasone 20 mg/day on days 1, 2, 8, 9, 15, 16, 22, and 23, until progression of disease, unacceptable toxicity, or for 24 cycles, whichever occurred first.
Period: Overall Study
Arm/Group | Oprozomib 150 mg 5/14 + Lenalidomide + Dexamethasone | Oprozomib 180 mg 5/14 + Lenalidomide + Dexamethasone | Oprozomib 210 mg 5/14 + Lenalidomide + Dexamethasone | Oprozomib 210 mg 2/7 + Lenalidomide + Dexamethasone | Oprozomib 240 mg 2/7 + Lenalidomide + Dexamethasone | Oprozomib 210 mg 2/7 + Cyclophosphamide + Dexamethasone
Started | 3 | 7 | 3 | 3 | 2 | 3
Completed | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 7 | 3 | 3 | 2 | 3
Not completed — Withdrawal by Subject | 0 | 2 | 1 | 0 | 1 | 1
Not completed — Study Terminated by Sponsor | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Other | 3 | 5 | 2 | 3 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oprozomib 150 mg 5/14 + Lenalidomide + Dexamethasone | Oprozomib 180 mg 5/14 + Lenalidomide + Dexamethasone | Oprozomib 210 mg 5/14 + Lenalidomide + Dexamethasone | Oprozomib 210 mg 2/7 + Lenalidomide + Dexamethasone | Oprozomib 240 mg 2/7 + Lenalidomide + Dexamethasone | Oprozomib 210 mg 2/7 + Cyclophosphamide + Dexamethasone | Total
Number analyzed (Participants) | 3 | 7 | 3 | 3 | 2 | 3 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.3 (6.1) | 68.9 (8.7) | 64.7 (2.5) | 64.7 (11.0) | 60.0 (5.7) | 67.7 (4.2) | 67.1 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 2 | 0 | 2 | 0 | 6
  Male | 3 | 5 | 1 | 3 | 0 | 3 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Not Hispanic or Latino | 3 | 6 | 3 | 3 | 2 | 3 | 20
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 3 | 5 | 3 | 2 | 2 | 3 | 18
  Other | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Reported | 0 | 1 | 0 | 0 | 0 | 0 | 1
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — A scale to assess a patient's disease status. 0 = Fully active, able to carry out all pre-disease performance without restriction;
  1. = Restricted in physically strenuous activity, ambulatory and able to carry out work of a light nature;
  2. = Ambulatory and capable of all self-care, unable to carry out any work activities. Up and about > 50% of waking hours;
  3. = Capable of only limited self-care, confined to bed or chair > 50% of waking hours;
  4. = Completely disabled, confined to bed or chair;
  5. = Dead.
  Participants
    Grade 0 (Fully active) | 1 | 4 | 3 | 1 | 1 | 3 | 13
    Grade 1 (Restricted but ambulatory) | 2 | 3 | 0 | 2 | 1 | 0 | 8
    Grade 2 (Ambulatory but unable to work) | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose-Limiting Toxicities (DLTs)
Description: DLTs were assessed according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.03. A DLT is defined as any of the following treatment-related events:
  * Any ≥ Grade 3 nonhematologic toxicity with the following conditions:
    * ≥ Grade 3 nausea, vomiting, diarrhea, or constipation only if for > 7 days despite optimal supportive care
    * Asymptomatic Grade 3 hypophosphatemia, Grade 3 hyperglycemia or toxicity solely due to dexamethasone, ≥ Grade 3 rash attributed to lenalidomide, and Grade 3 fatigue for < 14 days were not considered DLTs
  * Grade 4 neutropenia: absolute neutrophil count (ANC) < 0.5 × 10^9/L lasting ≥ 7 days, despite myeloid growth factor support
  * Febrile neutropenia
  * Grade 4 thrombocytopenia for ≥ 7 days or < 7 days with ≥ Grade 2 clinically significant bleeding or < 10,000 platelets requiring platelet transfusion, or Grade ≥ 3 with clinically significant bleeding or requiring platelet transfusion.
Time Frame: Cycle 1, 28 days
Population: All enrolled participants who received at least 1 dose of any study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Oprozomib 150 mg 5/14 + Lenalidomide + Dexamethasone | Oprozomib 180 mg 5/14 + Lenalidomide + Dexamethasone | Oprozomib 210 mg 5/14 + Lenalidomide + Dexamethasone | Oprozomib 210 mg 2/7 + Lenalidomide + Dexamethasone | Oprozomib 240 mg 2/7 + Lenalidomide + Dexamethasone | Oprozomib 210 mg 2/7 + Cyclophosphamide + Dexamethasone
Number analyzed (Participants) | 3 | 7 | 3 | 3 | 2 | 3
Participants | 2 | 2 | 2 | 0 | 1 | 0

2. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (AEs)
Description: Adverse events (AEs) were graded using NCI-CTCAE (version 4.03) and according to the following: Grade 1 = mild AE, Grade 2 = Moderate AE, Grade 3 = a severe AE, Grade 4 = life-threatening AE, and Grade 5 = death due to AE.
  A serious AE is an event that met 1 or more of the following criteria:
  * Death
  * Life-threatening experience
  * Required inpatient hospitalization or prolongation of an existing hospitalization
  * Resulted in persistent or significant disability/incapacity
  * A congenital anomaly birth defect in the offspring of an exposed female subject or offspring of a female partner of a male subject
  * Important medical events that, based upon appropriate medical judgment, jeopardized the participant and may have required medical or surgical intervention to prevent an outcome listed above.
  Treatment-related AEs are those considered related to at least 1 study drug by the investigator.
Time Frame: From first dose of any study treatment to 30 days after last dose; median duration of treatment was 29.1, 12.4, 11.3, 66.6, 7.8, and 46.4 weeks in each treatment group, respectively.
Population: Participants who received at least 1 dose of any study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Oprozomib 150 mg 5/14 + Lenalidomide + Dexamethasone | Oprozomib 180 mg 5/14 + Lenalidomide + Dexamethasone | Oprozomib 210 mg 5/14 + Lenalidomide + Dexamethasone | Oprozomib 210 mg 2/7 + Lenalidomide + Dexamethasone | Oprozomib 240 mg 2/7 + Lenalidomide + Dexamethasone | Oprozomib 210 mg 2/7 + Cyclophosphamide + Dexamethasone
Number analyzed (Participants) | 3 | 7 | 3 | 3 | 2 | 3
Participants
  Any treatment-emergent adverse event (TEAE) | 3 | 7 | 3 | 3 | 2 | 3
  TEAE ≥ grade 3 | 3 | 6 | 3 | 3 | 2 | 2
  Serious adverse events | 2 | 4 | 3 | 2 | 1 | 1
  TEAEs leading to discontinuation of study drug | 1 | 1 | 2 | 1 | 1 | 0
  Fatal adverse events | 0 | 0 | 0 | 0 | 0 | 0
  Treatment-related adverse events (TRAE) | 3 | 7 | 3 | 3 | 2 | 3
  TRAE ≥ grade 3 | 3 | 6 | 2 | 2 | 2 | 2
  Treatment-related serious adverse events | 2 | 4 | 2 | 1 | 1 | 1
  TRAEs leading to discontinuation of study drug | 1 | 1 | 2 | 1 | 1 | 0

3. Secondary Outcome: Plasma Oprozomib Concentration
Description: Plasma samples for oprozomib concentration assays were only collected for participants in the 5/14 dosing schedule groups.
  Oprozomib plasma concentrations were determined using liquid chromatography with tandem mass spectrometry.
Time Frame: Cycle 1 day 1 at 1 to 2.5 hours and 2.75 to 5 hours after end of infusion (EOI) and cycle 3 day 1 at predose and 1 to 2.5 hours and 2.75 to 5 hours after EOI.
Population: Participants in the 5/14 dosing schedule groups with available concentration data
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Oprozomib 150 mg 5/14 + Lenalidomide + Dexamethasone | Oprozomib 180 mg 5/14 + Lenalidomide + Dexamethasone | Oprozomib 210 mg 5/14 + Lenalidomide + Dexamethasone
Number analyzed (Participants) | 2 | 4 | 3
ng/mL
  Cycle 1 day 1, 1 - 2.5 hours post EOI: number analyzed (Participants) | 2 | 3 | 3
  Cycle 1 day 1, 1 - 2.5 hours post EOI | 497 (NA) — Standard deviation not calculated when N ≤ 2 | 632 (657) | 697 (435)
  Cycle 1 day 1, 2.75 - 5 hours post EOI: number analyzed (Participants) | 2 | 2 | 3
  Cycle 1 day 1, 2.75 - 5 hours post EOI | 299 (NA) — Standard deviation not calculated when N ≤ 2 | 15.8 (NA) — Standard deviation not calculated when N ≤ 2 | 78.0 (48.9)
  Cycle 3 day 1, predose: number analyzed (Participants) | 1 | 4 | 2
  Cycle 3 day 1, predose | 0.0 | 142 (285) | 0.0 (NA) — Standard deviation not calculated when N ≤ 2
  Cycle 3 day 1, 1 - 2.5 hours post EOI: number analyzed (Participants) | 1 | 4 | 2
  Cycle 3 day 1, 1 - 2.5 hours post EOI | 111 (NA) — Standard deviation not calculated when N ≤ 2 | 175 (303) | 178 (NA) — Standard deviation not calculated when N ≤ 2
  Cycle 3 day 1, 2.75 - 5 hours post EOI: number analyzed (Participants) | 1 | 4 | 2
  Cycle 3 day 1, 2.75 - 5 hours post EOI | 2.00 (NA) — Standard deviation not calculated when N ≤ 2 | 255 (323) | 69.1 (NA) — Standard deviation not calculated when N ≤ 2

4. Secondary Outcome: Overall Response Rate (ORR)
Description: ORR is defined as the percentage of participants with a best overall response of partial response (PR), very good PR (VGPR), complete response (CR), or stringent CR (sCR) based on the International Myeloma Working Group Uniform Response Criteria.
  PR: ≥ 50% reduction of serum M-protein and ≥ 90% reduction in urine M-protein or to < 200 mg/24 hrs, or a ≥ 50% decrease in dFLC. A ≥ 50% decrease in the size of soft tissue plasmacytomas present at baseline.
  VGPR: Serum and urine M-protein detectable by immunofixation but not electrophoresis or ≥ 90% decrease in serum M-protein with urine M-protein <100 mg/24 hrs. If disease measurable only by SFLC, ≥ 90% decrease in the difference between involved and uninvolved FLC levels (dFLC).
  CR: No immunofixation on serum and urine, disappearance of soft tissue plasmacytomas and <5% plasma cells in BM. Normal serum free light chain (SFLC) ratio if disease measurable only by SFLC.
  sCR: As for CR, and absence of clonal plasma cells in bone marrow (BM).
Time Frame: Disease response was assessed every 4 weeks for 24 cycles then every 8 weeks until end of treatment; median duration of treatment at the analysis cutoff date of 18 July 2016 was 29.1, 12.4, 11.3, 66.6, 7.8 and 46.4 weeks in each group, respectively
Population: All participants who received at least 1 dose of any study treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Oprozomib 150 mg 5/14 + Lenalidomide + Dexamethasone | Oprozomib 180 mg 5/14 + Lenalidomide + Dexamethasone | Oprozomib 210 mg 5/14 + Lenalidomide + Dexamethasone | Oprozomib 210 mg 2/7 + Lenalidomide + Dexamethasone | Oprozomib 240 mg 2/7 + Lenalidomide + Dexamethasone | Oprozomib 210 mg 2/7 + Cyclophosphamide + Dexamethasone
Number analyzed (Participants) | 3 | 7 | 3 | 3 | 2 | 3
percentage of participants | 66.7 [9.4 to 99.2] | 57.1 [18.4 to 90.1] | 66.7 [9.4 to 99.2] | 100.0 [29.2 to 100.0] | 50.0 [1.3 to 98.7] | 100.0 [29.2 to 100.0]

5. Secondary Outcome: Duration of Response (DOR)
Description: Duration of response was defined as the time from first evidence of partial response (PR) or better to confirmation of disease progression or death due to any cause.
  Median DOR was estimated using Kaplan-Meier methods. Participants who started a new anticancer therapy before documentation of disease progression or death, or who were alive without documentation of disease progression before the data cut-off date or who died or had disease progression immediately after more than 1 consecutively missed disease assessment visit were censored at the date of last disease assessment.
Time Frame: Disease response was assessed every 4 weeks for 24 cycles then every 8 weeks until end of treatment; median time on follow-up at the analysis cut-off date of 18 July 2016 was 14.1, 3.5, 2.6, 16.0, 3.6, and 11.2 months in each group, respectively.
Population: Participants who received at least 1 dose of any study treatment and who achieved a best overall response of sCR, CR, VGPR, or PR.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Oprozomib 150 mg 5/14 + Lenalidomide + Dexamethasone | Oprozomib 180 mg 5/14 + Lenalidomide + Dexamethasone | Oprozomib 210 mg 5/14 + Lenalidomide + Dexamethasone | Oprozomib 210 mg 2/7 + Lenalidomide + Dexamethasone | Oprozomib 240 mg 2/7 + Lenalidomide + Dexamethasone | Oprozomib 210 mg 2/7 + Cyclophosphamide + Dexamethasone
Number analyzed (Participants) | 2 | 4 | 2 | 3 | 1 | 3
months | NA [NA to NA] — Could not be estimated due to the low number of events | NA [NA to NA] — Could not be estimated due to the low number of events | NA [NA to NA] — Could not be estimated due to the low number of events | NA [NA to NA] — Could not be estimated due to the low number of events | NA [NA to NA] — Could not be estimated due to the low number of events | NA [NA to NA] — Could not be estimated due to the low number of events

6. Secondary Outcome: Progression-Free Survival (PFS)
Description: Progression-free survival is defined as the time from the start of treatment to disease progression or death (due to any cause), whichever occurred first. Median PFS was estimated using Kaplan-Meier methods. Participants who started a new anticancer therapy before documentation of disease progression or death, or who were alive without documentation of disease progression before the data cut-off date or who died or had disease progression immediately after more than 1 consecutively missed disease assessment visit were censored at the date of last disease assessment.
Time Frame: From first dose of study drug through the data cut-off date of 18 July 2016; median time on follow-up was 14.1, 3.5, 2.6, 16.0, 3.6, and 11.2 months in each group, respectively
Population: All participants who received at least 1 dose of any study treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Oprozomib 150 mg 5/14 + Lenalidomide + Dexamethasone | Oprozomib 180 mg 5/14 + Lenalidomide + Dexamethasone | Oprozomib 210 mg 5/14 + Lenalidomide + Dexamethasone | Oprozomib 210 mg 2/7 + Lenalidomide + Dexamethasone | Oprozomib 240 mg 2/7 + Lenalidomide + Dexamethasone | Oprozomib 210 mg 2/7 + Cyclophosphamide + Dexamethasone
Number analyzed (Participants) | 3 | 7 | 3 | 3 | 2 | 3
months | NA [NA to NA] — Could not be estimated due to the low number of events | NA [NA to NA] — Could not be estimated due to the low number of events | NA [NA to NA] — Could not be estimated due to the low number of events | NA [NA to NA] — Could not be estimated due to the low number of events | NA [NA to NA] — Could not be estimated due to the low number of events | NA [NA to NA] — Could not be estimated due to the low number of events

ADVERSE EVENTS:
Time Frame: From enrollment (for all-cause mortality) or from first dose of any study treatment (for adverse events) to 30 days after last dose; median duration of treatment was 29.14, 12.43, 11.29, 66.57, 7.79, and 46.43 weeks in each treatment group, respectively.
Arm/Group | Oprozomib 150 mg 5/14 + Lenalidomide + Dexamethasone | Oprozomib 180 mg 5/14 + Lenalidomide + Dexamethasone | Oprozomib 210 mg 5/14 + Lenalidomide + Dexamethasone | Oprozomib 210 mg 2/7 + Lenalidomide + Dexamethasone | Oprozomib 240 mg 2/7 + Lenalidomide + Dexamethasone | Oprozomib 210 mg 2/7 + Cyclophosphamide + Dexamethasone
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/7 | 0/3 | 0/3 | 0/2 | 0/3
Serious Adverse Events (participants affected / at risk) | 2/3 | 4/7 | 3/3 | 2/3 | 1/2 | 1/3
Other Adverse Events (participants affected / at risk) | 3/3 | 7/7 | 3/3 | 3/3 | 2/2 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Oprozomib 150 mg 5/14 + Lenalidomide + Dexamethasone (N=3) | Oprozomib 180 mg 5/14 + Lenalidomide + Dexamethasone (N=7) | Oprozomib 210 mg 5/14 + Lenalidomide + Dexamethasone (N=3) | Oprozomib 210 mg 2/7 + Lenalidomide + Dexamethasone (N=3) | Oprozomib 240 mg 2/7 + Lenalidomide + Dexamethasone (N=2) | Oprozomib 210 mg 2/7 + Cyclophosphamide + Dexamethasone (N=3)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Disease progression (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Bacterial sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Lung infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Neutropenic infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Neutropenic sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Myoclonus (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 2 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 0
Capillary leak syndrome (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 1 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Oprozomib 150 mg 5/14 + Lenalidomide + Dexamethasone (N=3) | Oprozomib 180 mg 5/14 + Lenalidomide + Dexamethasone (N=7) | Oprozomib 210 mg 5/14 + Lenalidomide + Dexamethasone (N=3) | Oprozomib 210 mg 2/7 + Lenalidomide + Dexamethasone (N=3) | Oprozomib 240 mg 2/7 + Lenalidomide + Dexamethasone (N=2) | Oprozomib 210 mg 2/7 + Cyclophosphamide + Dexamethasone (N=3)
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 1 | 2 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 2 | 1 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 2
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0
Dry eye (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 1 | 0 | 2 | 0 | 2
Abdominal distension (Gastrointestinal disorders) | 0 | 2 | 0 | 2 | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Cheilitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 4 | 1 | 2 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 5 | 3 | 3 | 1 | 2
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 3 | 0 | 1
Faecaloma (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Gastrointestinal toxicity (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0 | 2 | 0 | 0
Melaena (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 3 | 6 | 2 | 3 | 2 | 2
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 3 | 2 | 3 | 1 | 0
Asthenia (General disorders) | 0 | 2 | 0 | 1 | 0 | 1
Chills (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 2 | 4 | 1 | 3 | 1 | 1
Gait disturbance (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Oedema (General disorders) | 1 | 0 | 0 | 0 | 0 | 1
Oedema peripheral (General disorders) | 1 | 1 | 1 | 0 | 0 | 1
Pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Peripheral swelling (General disorders) | 1 | 1 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 2 | 0 | 1 | 0 | 1 | 0
Thirst (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Xerosis (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Candida infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Folliculitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Tinea infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 2
Urinary tract infection (Infections and infestations) | 1 | 1 | 0 | 1 | 0 | 0
Viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Compression fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 1
Aspartate aminotransferase decreased (Investigations) | 0 | 0 | 1 | 2 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0 | 0 | 1 | 0
Blood alkaline phosphatase decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Blood bicarbonate decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Blood bilirubin increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Blood chloride increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 1 | 0 | 1 | 0 | 0
Blood lactate dehydrogenase decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 1 | 0 | 1 | 0 | 0 | 0
Blood phosphorus increased (Investigations) | 0 | 0 | 0 | 2 | 0 | 0
Blood pressure increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Blood urea increased (Investigations) | 1 | 0 | 0 | 1 | 0 | 0
Blood uric acid decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Carbon dioxide increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 2 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 2 | 0 | 0
Neutrophil count increased (Investigations) | 0 | 0 | 0 | 2 | 0 | 0
Protein total decreased (Investigations) | 0 | 0 | 0 | 2 | 0 | 0
Red blood cell count decreased (Investigations) | 0 | 0 | 1 | 1 | 0 | 0
Weight decreased (Investigations) | 1 | 0 | 1 | 1 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 2 | 0 | 0
White blood cell count increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Appetite disorder (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 3 | 0 | 2 | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 2 | 0 | 0
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 2 | 1 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 2 | 1 | 0 | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 2 | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Coccydynia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 2 | 0 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 1 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 2 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 2 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Polycythaemia vera (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Burning sensation (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 4 | 2 | 2 | 1 | 2
Dizziness postural (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Dysgeusia (Nervous system disorders) | 1 | 0 | 2 | 2 | 1 | 1
Headache (Nervous system disorders) | 1 | 1 | 0 | 1 | 0 | 2
Hypoaesthesia (Nervous system disorders) | 1 | 1 | 0 | 1 | 0 | 0
Memory impairment (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 1 | 0 | 1 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 1 | 2 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Presyncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 1 | 0 | 3 | 0 | 0
Claustrophobia (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
Depressed mood (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 1 | 0 | 2 | 1 | 0
Irritability (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0
Sleep disorder (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 1 | 1 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Polyuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0 | 1 | 0 | 0
Genital rash (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 3 | 2 | 1
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 3 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 1 | 0 | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 2 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 1 | 0 | 1
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Aortic arteriosclerosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1 | 1 | 0
Hypotension (Vascular disorders) | 1 | 1 | 1 | 1 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2014-10-15): https://cdn.clinicaltrials.gov/large-docs/89/NCT01881789/Prot_000.pdf
  • Statistical Analysis Plan (2016-08-23): https://cdn.clinicaltrials.gov/large-docs/89/NCT01881789/SAP_001.pdf